CLINICAL TRIAL: NCT01242137
Title: Pharmacogenetic Effect on the Pharmacodynamics of Glibenclamide
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Assaf Harofe Medical Center, Assaf Harofe Medical Center
Other Study IDs: 169/09
Record Dates: First submitted 2010-11-14; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Extensive metabolizers
- Intermediate mtabolizers
- Poor metabolizers

SUMMARY:
Glibenclamide is metabolized by the hepatic enzyme P450 CYP2C9 to less active form. Polymorphism of this enzyme demonstrated clinical significance when examined on other drugs from the sulfonylurea drug family, to whom Glibenclamide is included.

The investigators assumption is that patients with less active alleles of the enzyme may show lower dose requirements of the drug for glycemic control, when compared to patients homozygotes to wild-type alleles.

ELIGIBILITY:
Inclusion Criteria:

* Tx with metformin and glibenclamide

Exclusion Criteria:

* Tx which affecting the P450 2C9 action
* Renal failure

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes type 2 patients treated with metformin and glibenclamide.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-10

PRIMARY OUTCOMES:
HbA1c | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe Medical Center, Beer Yakov, Israel